CLINICAL TRIAL: NCT06754761
Title: A Phase I, Open-label Study to Assess the Absolute Bioavailability of Ceralasertib (AZD6738) and Absorption, Distribution, Metabolism, and Excretion (ADME) of [14C]-Ceralasertib in Patients With Non-small Cell Lung Cancer, Ovarian Cancer, or Endometrial Cancer
Brief Title: Human ADME Study of [14C]-Ceralasertib (AZD6738) and Absolute Bioavailability of Ceralasertib
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D533BC00002
Record Dates: First submitted 2024-11-04; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Neoplasm
Keywords: non-small cell lung cancer; ovarian cancer; endometrial cancer; hADME, bioavailability; AZD6738; ceralasertib
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Endometrial Neoplasms | interventions — ceralasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary Treatment Arm - AZD6738 (Experimental): Part A - oral dose of Ceralasertib and a radiolabelled IV microdose of [14C]-Ceralasertib Part B - oral dose of [14C]-Ceralasertib
  Interventions: Drug: [14C] AZD6738; Drug: AZD6738 / ceralasertib

INTERVENTIONS:
Drug: [14C] AZD6738 — radiolabeled AZD6738 / ceralasertib
Drug: AZD6738 / ceralasertib — Ceralasertib (AZD6738) is a potent, selective inhibitor of the serine/threonine-specific protein kinase ATR

SUMMARY:
This is an open-label, two-part study in participants with NSCLC, ovarian cancer, or endometrial cancer and will be conducted at multiple study sites.

Participants will be assessed for study eligibility prior to admission to the study site.

Part A will assess the absolute bioavailability, determine the excretory routes of [14C]-Ceralasertib, and evaluate the PK parameters of a Ceralasertib oral dose and a radiolabelled IV microdose of [14C]-Ceralasertib.

Participants will be admitted to the study site pre-dose Part A and will remain at the study site for excreta (urine and faeces) collections, PK sampling and safety assessments. A washout period days will be observed between dosing in Part A and Part B. Part B will assess the ADME of [14C]-Ceralasertib.

Participants will be readmitted to the study site for Part B and will remain at the study site for excreta (urine, faeces, and any vomitus) collections, PK sampling, and safety assessments.

Participants will return to the study site for a Follow-up Visit after the last dose of Ceralasertib which will include routine safety assessments.

After the completion of Parts A and B, and following the Follow-up Visit, participants may be allowed further access to Ceralasertib if in the opinion of the investigator and medical monitor they may derive clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Participants are eligible to be included in the study only if all of the following criteria apply:

Age

1. Male or female ≥ 18 years of age (or the legal age of consent in the jurisdiction in which the study is taking place), at the time of signing the ICF.

   Type of Participant and Disease Characteristics
2. Sufficient ECOG performance status, life expectancy, and ability to swallow and retain oral medication
3. Adequate organ and marrow function
4. Willingness and ability to comply with study and follow-up procedures.
5. Able and willing to stay in hospital for specified residential periods following administration of Ceralasertib/[14C]-Ceralasertib
6. Regular bowel movements
7. Participants with NSCLC must have appropriately documented NSCLC diagnosis, mutation status, treatment history, and disease status according to protocol-specified eligibility criteria
8. Participants with Ovarian cancer must have appropriately documented ovarian cancer diagnosis, mutation status, treatment history, and disease status according to protocol-specified eligibility criteria 9. Participants with Endometrial cancer must have appropriately documented endometrial cancer diagnosis, treatment history, and disease status according to protocol-specified eligibility criteria 10. Sex and Contraceptive/Barrier Requirements: Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies 11. Informed Consent: patient must be capable of giving signed informed consent as described in Appendix A which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

* Participants are excluded from the study if any of the following criteria apply:

  1. History of Diagnosis of protocol-specified medical conditions
  2. Spinal cord compression or brain metastasis prior to start of study intervention unless asymptomatic and stable
  3. Persistent toxicities (CTCAE Grade ≥ 2), with the exception of alopecia and vitiligo, caused by previous anticancer therapy.
  4. History of allogenic organ transplant or autoimmune or inflammatory disorders requiring use of immunosuppressive medications with some protocol specified conditions/exceptions
  5. Any medical or surgical condition that would preclude adequate absorption of Ceralasertib
  6. Inadequate cardiac function / status or other cardiovascular diseases
  7. Participants with active infection requiring systemic antibiotics, antifungal or antiviral drugs
  8. Any evidence of severe or uncontrolled systemic disease, as judged by the investigator that would make it undesirable for the participant to participate in the study or would jeopardise compliance with the protocol
  9. Protocol-specified prior/concomitant therapy exclusions
  10. Protocol-specified prior/concurrent clinical study experience
  11. Other Exclusions including but not limited to tobacco/nicotine and/or alcohol use, or drug/alcohol abuse history
  12. Not currently pregnant, breast-feeding, or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-01-17 (Estimated); Primary Completion 2025-08-08 (Estimated); Study Completion 2025-08-08 (Estimated)

PRIMARY OUTCOMES:
To evaluate absolute bioavailability Ceralasertib and PK of Ceralasertib and [14C]-Ceralasertib after administration of oral dose of Ceralasertib and IV [14C]-Ceralasertib (Part A | Through end of Part A, approximately 5 weeks including screening period
  Absolute bioavailability (F) of Ceralasertib and PK parameters
To determine the rates and major excretory routes of Ceralasertib and its metabolites after IV dose of [14C]-Ceralasertib (Part A) and a oral dose of [14C]-Ceralasertib (Part B) | Through end of Part B, approximately 10 weeks including screening period
  [14C]-Ceralasertib (Part A) or total radioactivity (Part B) recovery in urine and faeces
To characterise the PK of Ceralasertib and total radioactivity following oral dose of [14C]-Ceralasertib including the extent of distribution into blood cells (Part B) | Through end of the part B, approximately 10 weeks (Including screening period)
  AUCinf
To characterise the PK of Ceralasertib and total radioactivity following oral dose of [14C]-Ceralasertib including the extent of distribution into blood cells (Part B) | Through end of the part B, approximately 10 weeks (Including screening period)
  AUClast
To characterise the PK of Ceralasertib and total radioactivity following oral dose of [14C]-Ceralasertib including the extent of distribution into blood cells (Part B) | Through end of the part B, approximately 10 weeks (Including screening period)
  Cmax
To characterise the PK of Ceralasertib and total radioactivity following oral dose of [14C]-Ceralasertib including the extent of distribution into blood cells (Part B) | Through end of the part B, approximately 10 weeks (Including screening period)
  tmax
To characterise the PK of Ceralasertib and total radioactivity following oral dose of [14C]-Ceralasertib including the extent of distribution into blood cells (Part B) | Through end of the part B, approximately 10 weeks (Including screening period)
  t1/2(lambda)z
To characterise the PK of Ceralasertib and total radioactivity following oral dose of [14C]-Ceralasertib including the extent of distribution into blood cells (Part B) | Through end of the part B, approximately 10 weeks (Including screening period)
  Ratio of AUCinf of plasma Ceralasertib relative to AUCinf of plasma total radioactivity
To characterise the PK of Ceralasertib and total radioactivity following oral dose of [14C]-Ceralasertib including the extent of distribution into blood cells (Part B) | Through end of the part B, approximately 10 weeks (Including screening period)
  Ratio of AUCinf of whole blood total radioactivity relative to AUCinf of plasma total radioactivity
To characterise the PK of Ceralasertib and total radioactivity following oral dose of [14C]-Ceralasertib including the extent of distribution into blood cells (Part B) | Through end of the part B, approximately 10 weeks (Including screening period)
  Pharmacokinetic activity of ceralasertib present in urine

SECONDARY OUTCOMES:
To provide biologic samples for metabolic profiling and identification after oral dose of [14C]-Ceralasertib (Part B) | Through end of the part B, approximately 10 weeks (Including screening period)
  Quantification and identification of major metabolites of Ceralasertib in plasma and excreta (will be reported separately)
To assess the safety of Ceralasertib in participants with NSCLC, ovarian cancer, or endometrial cancer (Parts A and B) | Through study completion, approximately 9 - 11 weeks, with screening included
  Incidence and severity of AEs Incidence of laboratory abnormalities, based on haematology, clinical chemistry, and urinalysis test results 12-lead ECG parameters Vital signs measurements Physical examinations

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Research Site, Liverpool
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/